CLINICAL TRIAL: NCT07304375
Title: Effects of Aerobic Exercise and Daytime Sleep on Neurorehabilitation and Functional Abilities in Multiple Sclerosis: Evidence of Training the Brain in Neurorehabilitation
Brief Title: Effects of Exercise and Sleep on Motor Learning and Functional Abilities in Multiple Sclerosis
Acronym: ExSiMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Martin Ballegaard MD PhD, Clinical Associate Professor, Zealand University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SJ-1040; SJ-1040 (Other: De Videnskabelige Komitéer)
Record Dates: First submitted 2025-11-26; First posted 2025-12-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Exercise; Sleep; Motor Learning; Memory; Multiple Sclerosis
Keywords: Aerobic Exercise; Daytime Sleep; Sleep; Learning Ability; Motor Learning; Memory; Cognitive Function; Neurorehabilitation
MeSH Terms: conditions — Motor Activity; Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Due to large between-patient variability of motor function, the participants will have more than one intervention with a wash-out period in between and with a change in task complexity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise - GXT (Experimental): The aerobic exercise will consist of about 20 minutes of Graded Exercise Training (GXT) on an ergometer bike. The experimenter will instruct and motivate the participant through the aerobic exercise.
  Interventions: Other: Aerobic Exercise
- Control - Rest (No Intervention): The participant will rest in a sitting position in a quiet room for 20 minutes. The participant is allowed to read or engage in similar quiet and sitting activities.
- Daytime Sleep - Nap (Experimental): The participants will be asked to try and take a 30-minute nap. The participant will be provided with a bed in a dark and quiet room.
  Interventions: Behavioral: Daytime Sleep - Nap

INTERVENTIONS:
Other: Aerobic Exercise — The Aerobic Exercise Intervention consists of 20 minutes of Graded Exercise Test (GXT) on an ergometer bike. The participants start with 5 minutes of warm-up. The wattload will then be increased until exhaustion.
  Arms: Aerobic Exercise - GXT
Behavioral: Daytime Sleep - Nap — The Daytime sleep consists of a 30-minute nap after the acquisition of the visuomotor accuracy tracking task. The participants will be asked to rest in a supine position in a bed in a dark and quiet room.
  Arms: Daytime Sleep - Nap

SUMMARY:
The ExSiMS study is a randomized, controlled crossover study including 20 individuals (18-70 years) diagnosed with relapsing remitting Multiple Sclerosis (MS) This project investigates, through behavioral and neurophysiological measurements, how aerobic exercise on an ergometer bike and sleep in the form of a nap and overnight sleep may enhance cortical motor skill learning evaluated by a complex hand motor skill test and thereby improve functional capacity in individuals with MS. Beyond the effect on motor skill learning, the project investigate the effect on electroencephalography (EEG) - electromyography (EMG) coherence.

The study hypothesizes that individuals with neurological conditions, such as multiple sclerosis (MS), may experience beneficial effects on specific motor rehabilitation through systematically planned cardiovascular exercise and sleep scheduling, due to positive impacts on memory consolidation.

Aims:

* Investigate the brain's neurophysiological responses and memory effects following a training intervention and, separately, sleep, in the form of a power nap, in individuals with MS.
* Examine whether these effects persist beyond the few days previously observed in healthy individuals by implementing a longer-term intervention.
* Explore whether the training effect is influenced by disease activity in the brain, such as during relapses and during immunosuppressive treatment.
* Assess whether the presence of abnormally reduced cognitive endurance (fatigue) affects the impact of the intervention involving exercise and sleep.

The study is based on documented positive effects of physical activity and sleep in both young and older adults, as well as in individuals recovering from stroke. The research thus offers promising perspectives for broader applications within neurorehabilitation, and particularly for MS, as the disease is associated with functional impairments. At the same time, both physical exercise and sleep represent meaningful interventions that should be thoughtfully integrated into rehabilitation strategies.

DETAILED DESCRIPTION:
The ExSiMS-project consists of both a proof-of-concept study and a longitudinal study.

In both studies, participants will perform a visuomotor accuracy tracking task (VATT) with their dominant hand on the main experimental days. The participants will wear EEG and EMG electrodes during the VATT. This will make it possible to investigate cortical activity during skill acquisition and later analyse the corticomuscular coherence. After the VATT, the participants will be randomized to either 20 min aerobic exercise on an ergometer bike, a short 30-minute nap or control (sitting rest). The interventions will run over a longer period of time in the longitudinal study.

The participants will be asked to do a retention test of the visuomotor accuracy tracking task 24 hours later.

The studies will run over more experiment days divided into two experiment blocks of at least two experiment days separated by between two weeks to three months.

Methods:

* Electroencephalography (EEG) and Electromyography (EMG)
* Actigraphy/Accelerometry
* Visuomotor Accuracy Tracking Task (VATT)
* Training on an Ergometerbike: Graded Exercise Test (GXT), High Intensity Interval Training (HIIT)
* Polysomnography (PSG)

ELIGIBILITY:
Inclusion Criteria:

* Competent individuals (aged 18-70) diagnosed with early relapsing-remitting MS
* Expanded Disability Status Score, 1 < EDSS < 4.5
* MRC muscle strength ≥ 4+ in the dominant hand

Exclusion Criteria:

* Implanted devices, such as pacemakers or stimulators
* Epilepsy or neuromuscular diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Motor/Skill Learning | Assessed on experiment days 1, 2, 3 and 4.
  Visuomotor accuracy tracking task. Online and offline effects. Unit: Range from 0 (lowest) to 100 (highest) percent.
Neurophysiological Measurement I - Cortical Activity | Assessed on experiment day 1, 2, 3 and 4.
  Cortical activity will be measured with electroencephalography (EEG) during skill acquisition. Unit: EEG Power in several frequency bands.
Neurophysiological Measurement II - Muscular Activity | Assessed on experiment day 1, 2, 3 and 4.
  Muscle activity will be measured with electromyography (EMG) during skill acquisition. Unit: EMG amplitude.
Neurophysiological Measurement III - Corticocortical Functional Connectivity | Assessed on experiment day 1, 2, 3 and 4.
  Corticocortical functional connectivity will me measured as functional coupling in EEG during skill acquisition. Unit: functional coupling in EEG (scale 0-1).
Neurophysiological Measurement IV - Corticomuscular Functional Connectivity | Assessed on experiment day 1, 2, 3 and 4.
  Corticomuscular functional connectivity during skill acquisition will be measured with functional coupling between EEG and EMG. Unit: functional coupling in EEG-EMG.
Neurophysiological Measurement V - Muscular Functional Connectivity | Assessed on experiment day 1, 2, 3 and 4.
  Muscular functional connectivity during skill acquisition will be assessed using EMG-EMG coherence between M. Abductor Pollicis Brevis and First Dorsal Interosseus. Unit: EMG-EMG coherence (0-1)

SECONDARY OUTCOMES:
Actigraphy | Assessment from day 0 to experiment day 4.
  Measurement of sedentary, moderate, and vigorous activity during the experiment period. Unit = hours:min.
Sleep quality - self reported sleep latency. | Assessed at the days leading up to experiment days 1,2,3, and 4.
  Self-reported sleep latency will be measured by the National Sleep Foundation Sleep Diary translated to Danish. Unit: Hour:minutes.
Sleep quality - Self reported sleep duration | Assessed at the days leading up to experiment days 1,2,3, and 4.
  Self-reported sleep duration will be measured by the National Sleep Foundation Sleep Diary translated to Danish. Unit: Hour:min.
Physical fitness level - work load | Assessed on either experiment day 1 or 3.
  Graded exercise test (GXT) on an ergometer bike - maximum work load. Unit: watt
Physical fitness level - heart rate | Assessed on either experiment day 1 or 3
  Graded exercise test (GXT) on an ergometer bike - heart rate measured with a chest strap. Unit: beats per minute (BPM).
Physical fitness level - rating of perceived exertion | Assessed on either experiment day 1 or 3.
  Graded exercise test (GXT) on an ergometer bike - rating of perceived exertion with the Borg scale. Unit: Borg scale 6-20 (6 = rest, 20 = maximal exhaustion).

OTHER OUTCOMES:
Wakefulness | Assessed on experiment days 1, 2, 3 and 4.
  Wakefulness will be measured by the Stanford Sleepiness Scale: From 1 to 7. 1= "Feeling active and vital; alert; wide awake". 7= "Almost in reverie; sleep onset soon; lost struggle to remain awake. X = Asleep".
Handedness | Assessed on day 0.
  Handedness questionnaire to determine the participant's dominant hand. Unit: Laterality index (-100.00 (lefthanded) to 100.00 (righthanded).
Reaction Time Task | Assessed on day 0.
  A simple Reaction Time Task on a computer. Unit: ms.
The fatigue scale for motor and cognitive functions (FSMC) | Assessed on day 0.
  Questionnaire measuring fatigue in individuals with Multiple Sclerosis. Unit: FSMC_total = Points from 20-100 (≥ 43 Mild Fatigue, ≥ 53 Moderate Fatigue, ≥ 63 Severe Fatigue).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ballegaard, Principal Investigator — Zealand University Hospital - Roskilde
Locations (2):
- Denmark (2):
  - Section of Movement and Neuroscience, Department of Nutrition, Exercise, and Sports, University of Copenhagen, Copenhagen
  - Zealand University Hospital Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: No